CLINICAL TRIAL: NCT04179435
Title: Développement Cognitif et cérébral Chez Les Adolescents Souffrants d'un Syndrome de Gilles de la Tourette
Brief Title: Cognitive and Brain Development in Adolescents With Gilles de la Tourette Syndrome
Acronym: CADETS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C19-11; 2019-A00992-55 (Registry Identifier: CADETS)
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Tourette Syndrome in Adolescence

STUDY DESIGN:
Intervention Model Description: Between group comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourette syndrome (Other): Patients with Tourette syndrome aged 13 - 18 y.o. Interventions : Brain scans, cognitive testing, TMS measures
  Interventions: Behavioral: Behavioral testing on cognitive computerized tasks; Other: brain MRI; Other: TMS
- Controls (Other): Controls matched to Tourette syndrome group nterventions : Brain scans, cognitive testing, TMS measures
  Interventions: Behavioral: Behavioral testing on cognitive computerized tasks; Other: brain MRI; Other: TMS

INTERVENTIONS:
Behavioral: Behavioral testing on cognitive computerized tasks — Testing on cognitive computerized tasks
Other: brain MRI — Brain MRI scans
Other: TMS — Measure of the cortical inhibitory capacity using TMS measures

SUMMARY:
In children with neurodevelopmental disorders, adolescence is usually associated with a reshaping of the clinical picture and symptomatology. Tourette syndrome (TS) is a paradigmal neurodevelopmental syndrome characterised by involuntary paroxysmal movements (motor tics) and vocalisation (vocal tics) often associated with various psychiatric disorders. The neuronal and cognitive mechanisms associated with TS symptoms improvement during adolescence, or the persistence in adulthood remains unknown, and this is what we aim to address in this study.

DETAILED DESCRIPTION:
Thus, the aims of the present project is threefold:

Aim 1: To evaluate the maturation of cognitive functions in adolescents with TS compared to typically developing adolescents.

To achieve this aim, three distinct cognitive dimensions will be assessed in all subjects (patients and controls): (i) reward sensitivity and habit formation; (ii) cognitive impulsivity and action control and (iii) self-agency.

Aim 2: To identify neuronal correlates of cognitive function and brain development in health and disease. To achieve this aim, we will use a combined behavioural (as described in Aim 1), (i) neuroimaging and (ii) TMS approaches.

Aim 3: To predict clinical outcome . In this part of the project we aim to identify behavioural, imaging or neurophysiological markers of clinical outcome in patients with TS.

ELIGIBILITY:
Inclusion Criteria:

* Tourette syndrome
* Ages 13 - 18
* Acceptance to perform the Brain MRI
* Acceptance to perform the cognitive testing
* Acceptance to perform the TMS measures

Exclusion Criteria:

* Learning disability
* Incompatibility with MRI procedure (metal body implants, pregnancy)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Behavioral test main outcome measures [1] | from 16 to 20 months
  reaction times
Behavioral test main outcome measures [2] | from 16 to 20 months
  discounting factor
Behavioral test main outcome measures [3] | from 16 to 20 months
  number of premature responses
Behavioral test main outcome measures [4] | from 16 to 20 months
  agency composite scores
Brain MRI scan measures | from 16 to 20 months
  whole brain structural connectivity, whole brain functional connectivity, brain cortical and subcortical structures volumes and morphology
Transcranial magnetic stimulation | from 16 to 20 months
  intracortical inhibition (SICI) scores

CONTACTS AND LOCATIONS:
Overall Officials: Worbe Yulia, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atkinson-Clement C, Duflot M, Lastennet E, Patsalides L, Wasserman E, Sartoris TM, Tarrano C, Rosso C, Burbaud P, Deniau E, Czernecki V, Roze E, Hartmann A, Worbe Y. How does Tourette syndrome impact adolescents' daily living? A text mining study. Eur Child Adolesc Psychiatry. 2023 Dec;32(12):2623-2635. doi: 10.1007/s00787-022-02116-1. Epub 2022 Dec 2. PMID 36460852